CLINICAL TRIAL: NCT05380921
Title: Testing a Novel Dry Electrode Headset for Electroencephalography Telehealth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: IIR 19-408; HX003107 (Other Grant/Funding Number: VA Merit Grant)
Record Dates: First submitted 2022-03-16; First posted 2022-05-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy
Keywords: EEG; epilepsy; electroencephalography; Point-of-Care Systems
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: study subjects will receive first a standard EEG study and then after this a dry electrode EEG study (in this sequence) at each study visit.
Who Masked: Outcomes Assessor
Masking Description: study investigators will score EEG quality in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- standard EEG (Experimental): all subjects will receive both a standard EEG and a dry electrode EEG
  Interventions: Device: standard EEG
- dry electrode EEG (Experimental): all subjects will receive both a standard EEG and a dry electrode EEG
  Interventions: Device: dry electrode EEG

INTERVENTIONS:
Device: standard EEG — all subjects will receive both a standard EEG and a dry electrode EEG
  Arms: standard EEG
Device: dry electrode EEG — all subjects will receive both a standard EEG and a dry electrode EEG
  Arms: dry electrode EEG

SUMMARY:
This study will improve access of Veterans with epilepsy living in rural areas to the most important diagnostic procedure for the care of patients with epilepsy: the routine electroencephalogram (EEG). The investigators will test a new method for recording EEG which uses a novel dry electrode system headset that does not require an EEG technologist to operate. The headset integrates the EEG electrodes and amplifier into a compact system which is easily placed on the head. This approach could make it possible for a nurse or nurse assistant with minimal training to record an EEG in a rural community based outpatient clinic (CBOC) as part of an epilepsy telemedicine outreach program along with clinical interviews. The investigators will compare performance of this dry electrode system to standard EEG when it is used by EEG technologists in three VA medical centers. This project has the potential to improve access of Veterans to the EEG procedure and decrease cost to the Veterans Health Care System.

DETAILED DESCRIPTION:
Title: Testing a Novel Dry Electrode Headset for Electroencephalography Telehealth

Justification: Many Veterans live far away from a VAMC with substantial electroencephalography (EEG) expertise. Travel is difficult for epilepsy patients since they often cannot drive. The investigators propose to study a novel dry electrode system (DES) which does not require EEG technologists to operate and can be operated by a nurse assistant. This DES integrates the electrodes and EEG amplifier into a compact headset which is easily placed on the head (without skin preparation) and could be used in an epilepsy telemedicine outreach program along with clinical interviews. The investigators have performed three preliminary studies with DES headsets. In the first two studies in 33 Veterans performed at a VAMC, the investigators found that the DES was quick to apply, taking only 5-6 minutes to put on by a research subject with the assistance of a neurologist. Subjects preferred the DES headset over the standard EEG system (SES). In the third study a nurse performed 30 DES recordings in a VA community based outpatient clinic (CBOC). Rating of the EEG recordings on a five point scale by three board certified clinical EEG experts (after automated EEG artifact reduction was applied to the recordings) showed that all 30 recordings were of acceptable quality (rated 3 out of 5 or higher with some artifact present) and 18 of 30 recordings were of good quality (rate 4 or above with only minor artifacts present).

Gaps to be address: This study will improve access of Veterans with epilepsy living in rural areas to the most important diagnostic procedure for the care of patients with epilepsy: the routine EEG. Being able to perform routine EEG in CBOCs can decrease cost to the VA system since DES EEG systems are less expensive and because Veterans will not have to travel to VAMCs for EEG. This study will also test the DES system to make sure it can record epileptiform transients (ETs), the pattern in EEG which indicates that patients have epilepsy.

Innovativeness: This study is innovative because it will use a new recording system for EEG that just got FDA approval. This new DES EEG recording system provides a method for recording EEG which is cheaper and much easier to perform than conventional EEG. This study is also innovative because it will test for the first time if a DES can reliably record ETs. (The FDA approval for the DES system was based on EEG signal quality only and not whether it could reliably detect ETs.) The study will also use a new FDA-approved method for automatically removing artifactual signals which can obscure DES EEG recordings.

Specific Aims: The first aim of the project is to test the ability of the DES to record ETs versus the SES. The second aim is to collect data on appointment wait time, appointment cancellation rate, and procedure cost of DES versus SES to project the improvement in Veteran access and potential cost-benefit of DES EEG performed in CBOCs versus SES EEG performed in VAMCs.

Project Methods: This is a diagnostic device trial which will be performed at three sites: the Charleston VAMC, Durham VAMC, and Miami VAMC. For Specific Aim 1, 400 Veterans (200 with a history of an abnormal EEGs in which ETs were recorded and 200 prospective Veterans scheduled for an outpatient EEG) will be recruited to have a DES EEG procedure and a SES EEG procedure performed during a single study visit in a VAMC by an EEG technologist. Each EEG recording will be interpreted and rated for technical quality by three study investigators, who will also annotate the location of ETs in each EEG recording. The fraction of EEGs which demonstrate ETs and the technical quality ratings will be compared. For Specific Aim 2, data will be collected on 300 prospective Veterans scheduled for an outpatient routine EEG, including appointment cancellation rate, travel cost, and other patient factors. Costs for EEG equipment/supplies as well as technician effort/salary and nurse and nurse assistant effort/salary will also be collected. This will be used to project the potential improvement in patient access and potential cost savings of a nurse or nurse technician performing outpatient DES EEG in a CBOC versus an EEG technician performing outpatient SES EEG in a VAMC.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1: subjects with history of an EEG within last five years at VA
* Aim 2: subjects scheduled for an outpatient EEG

Exclusion Criteria:

* weave hairstyles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Detection of epileptiform activity in EEG. | Through study completion, approximately 4 years.
  Measuring the technical quality of the DES to record ETs versus the SES.

SECONDARY OUTCOMES:
Procedure Costs of EEG. | Through study completion, approximately 4 years.
  Measuring procedure cost of DES versus SES.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Halford, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (3):
- United States (3):
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Richmond VA Medical Center, Richmond, VA, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Halford JJ, Campobello G, Brinkmann BH, Stead M, Rampp S, Remi J, Nilsen KB, Dauwels J, Galanti M, Dean BC, Winkler S, Ehrenberg JA, Pfaff J, Sullivan GJ. Letter to the Editor: Announcement of a Call for Proposals for biomedical waveform coding. Clin Neurophysiol. 2024 Sep;165:88-89. doi: 10.1016/j.clinph.2024.06.010. Epub 2024 Jul 2. No abstract available. PMID 38991377